CLINICAL TRIAL: NCT03310099
Title: Unsaturated Fatty Acids Enriched-diet to Improve Cardiorespiratory Fitness, Metabolic Flexibility and Glucose Tolerance in Obese Patients: a Feasibility Study
Brief Title: Unsaturated Fatty Acids Enriched-diet to Improve Cardiorespiratory Fitness, Metabolic Flexibility and Glucose Tolerance in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20011363
Record Dates: First submitted 2017-10-02; First posted 2017-10-16 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure With Normal Ejection Fraction; Obesity
Keywords: Obesity; Heart failure with preserved ejection fraction; HFpEF; unsaturated fatty acids; cardiorespiratory fitness; dietary intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention (Experimental): Dietary intervention aimed at increasing UFA consumption. The face-to-face intervention will be performed by a research nutritionist that reviews the dietary recall and provides a list of commonly available foods rich in unsaturated fatty acids (UFA) (monounsaturated [MUFA] and polyunsaturated fatty acids [PUFA]), together with individual instructions on how to integrate the recommended foods in the daily dietary pattern based on the dietary recall, and also to emphasize that the recommended food should be consumed as listed, and not as part of processed food (i.e., guacamole for avocado, hazelnut chocolate for nuts, pesto for olive oil, fish sticks for fatty fish). Extra-virgin olive oil or canola oil or nuts will be considered first choice for daily consumption of UFA-rich food, but a list of daily food substitutes will be also provided .
  Interventions: Behavioral: Increasing daily unsaturated fatty acid consumption

INTERVENTIONS:
Behavioral: Increasing daily unsaturated fatty acid consumption — Investigators will provide participant with detailed information about the consumption of food rich in unsaturated fatty acids (UFA) like extra-virgin olive oil, canola oil or mixed nuts, and they will provide specific recommendations based on the participant's diet. The investigators will follow up with a weekly phone call to assure that the dietary recommendations are clear and that the participants can integrate the suggestions into their daily diets.

SUMMARY:
The investigators hypothesize that a dietary intervention aimed at increasing unsaturated fatty acids (UFA) consumption is feasible and has the potential to improve cardiorespiratory fitness, metabolic flexibility and glucose tolerance in symptomatic obese heart failure with preserved ejection fraction (HFpEF) patients.

DETAILED DESCRIPTION:
Twelve obese HFpEF subjects with exercise intolerance (reduce cardiorespiratory fitness measured at maximal cardiopulmonary exercise test [CPX]) will be assigned to a single-arm open-label dietary intervention in which subjects are encouraged and financially supported to increase daily UFA consumption. The investigators will measure dietary compliance with a validated 24-hour dietary recall and with objective operator-independent biomarkers of UFA consumption.

The investigators will also measure the effects of UFA supplementation on: metabolic flexibility, glucose tolerance and body composition. Participants will have the option to participate in overnight session in the whole indirect calorimeter room (WIC) at baseline and at the end of the study.

ELIGIBILITY:
Major Inclusion Criteria:

* Body Mass Index (BMI) ≥30 kg/m2 (obesity) or total body fat percentage >25% in men and >35% in women
* A confirmed clinical diagnosis of stable HF (New York Heart Association [NYHA] class II-III) on maximally tolerated heart failure (HF) optimal medical regimen (without major changes in the prior month)
* Left Ventricular Ejection Fraction (LVEF)>50% documented in the prior 12 months

Major Exclusion Criteria:

* Concomitant conditions or treatment which would affect completion or interpretation of the study (i.e.,physical inability to walk or run on treadmill);
* Significant ischemic heart disease, angina, uncontrolled arterial hypertension, atrial fibrillation, moderate to severe valvular disease, chronic pulmonary disease, anemia (Hemoglobin<10 g/dL)
* Electrocardiography (ECG) changes (ischemia or arrhythmias) that limit maximum exertion during cardiopulmonary exercise test
* Comorbidity limiting survival
* Stage IV-V kidney disease (estimated Glomerular Filtration Rate<30)
* Fluid overload
* Pregnancy
* Current use of unsaturated fatty acids (UFA) supplement (i.e., omega-3).
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour dietary recall | Baseline to 12 weeks
  Measured with validated 24-hour dietary recall (non-self administered)
Change in dietary compliance (biomarkers) | Baseline to 12 weeks
  Measured by changes in biomarkers of unsaturated fatty acid consumption

SECONDARY OUTCOMES:
Change in metabolic flexibility | At baseline and 12 weeks
  Area under the curve change of respiratory quotient measured during overnight stay for 14 hours in the WIC
Change in body composition | At baseline and at 12 weeks
  Assessed by dual energy X-ray absorptiometry (DXA)
Change in glucose tolerance | At baseline and at 12 weeks
  Oral glucose tolerance test (OGTT) measures plasma glucose and insulin

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Carbone, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to present the data promptly upon analysis as an abstract to a national meeting and/or a manuscript.